CLINICAL TRIAL: NCT06024564
Title: Sonu Real-World Use Clinical Study to Treat Moderate to Severe Nasal Congestion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business/strategic decision
Sponsor: Third Wave Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-007
Record Dates: First submitted 2023-08-27; First posted 2023-09-06 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): Participants will receive Acoustic Resonance Therapy using the Sonu headband and App, twice a day, for 90 days
  Interventions: Device: Sonu Acoustic Resonance Therapy

INTERVENTIONS:
Device: Sonu Acoustic Resonance Therapy — Participants will receive Sonu treatment twice a day for 90 days

SUMMARY:
Real world utilization of Acoustic Resonance Therapy for symptoms of Nasal Congestion

DETAILED DESCRIPTION:
This is an interventional study designed to gather data on real world utilization of Acoustic Resonance Therapy for treating moderate to severe nasal congestion

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Present with symptoms of chronic nasal congestion
* Have a 24 hour reflective nasal congestion subscore of the TNSS of 2 or more on a 0 to 3 scale at the time of screening

Exclusion Criteria:

* Head, nasal or sinus surgery within 3 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Weekly Utilization-Frequency | 90 days
  Weekly utilization of Sonu treatment, measured as the frequency or number of times used per week
Weekly Utilization-Duration | 90 days
  Weekly utilization of Sonu treatment, measured as the duration of treatment received per week

SECONDARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 90 days
  24-hour TNSS; Minimum score=0 (no symptoms), Maximum score=12 (severe symptoms). Lower scores are better and reflect less symptoms.
Asthma Control | 90 days
  Asthma Control Test (ACT) Score; Minimum score = 5 (poor control of asthma). Maximum score = 25 (complete control of asthma). Higher scores reflect greater asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Johnson, MD, Principal Investigator — San Francisco Otolaryngology Medical Group
Locations (1):
- San Francisco Otolaryngology Medical Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No